CLINICAL TRIAL: NCT01700634
Title: fMRI Evaluation of Pain Central Sensitization Phenomena in Subjects With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Jordi Monfort, MD, Parc de Salut Mar
Other Study IDs: MON-SC-2012-01
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis
Keywords: fMRI, BOLD, pressure stimuli
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- OA patients with HIGH central sensitization: Central sensitization will be defined by the presence of both spreading sensitization and temporal summation to repeated pressure pain stimulation (Arendt-Nielsen et al. 2010, Graven-Nielsen et al. 2010, Woolf 2010, Imamura et al. 2008, Nijs et al. 2010).
- OA patients with LOW central sensitization
- Control subjects

SUMMARY:
The aim of this project is to investigate fMRI ability to identify pain central sensitization in chronic knee OA. Patients with high and low central sensitization and healthy control subjects will be included. Central sensitization will be clinically defined based on the evidence of regional spread of pain (spreading sensitization) and increased pain response to repeated stimulation (temporal summation). Operatively, a patient will be assigned to high sensitization group when showing (i) clinical evidence of pain or altered sensations spread beyond the knee joint by manual palpation, (ii) a minimum of 3 anatomical sites around the knee showing a pressure pain threshold below 4 kg/cm2 (tender points), (iii) pain score of 4 points or more in a 11-point scale during 4 kg/cm2 pressure stimulation on the anterior/medial surface of the tibial bone (the site selected for the fMRI experiment) and (iv) increase of at least 1 point in a 11-point scale after 10 repeated pressure stimulation on the tenderest point around the knee.

A three-step strategy is proposed to characterize the phenomenon by assessing (i) brain response to direct pressure stimulation on the painful knee, which will reflect the combination of peripheral and central sensitization; (ii) brain response to pressure stimulation on a non-arthritic hyperalgesic area (i.e., the anterior surface of the tibia), which will mostly reflect central sensitization mediated at the spinal cord level, and (iii) brain response to moderately painful heat stimulation on a healthy skin area (i.e., volar forearm), which will reflect central sensitization occurring in the brain and involving the highest-level pain modulatory mechanisms. An additional evaluation is proposed using resting-state fMRI to assess potential alterations in baseline brain functional organization.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  1. A diagnosis of knee OA and suitable for the study as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
  2. Have a radiological and clinical diagnosis of knee OA based upon American College of Rheumatology (ACR) criteria (1986) affecting at least one knee of a minimum of 3 months in symptom duration prior to screening.
  3. Subject is either male or female and at least 45 years of age.
  4. A minimum of 4 out of 10 on the numerical rating scale (Brief Pain Inventory- BPI item 5) at screening and/ or a requirement for the use of an analgesic for the pain in the OA knee. In addition, baseline pain must be stable for at least 72 hours prior to fMRI assessment or fMRI assessment may be delayed.
  5. A maximum of 8 out of 10 on the NRS at screening. Enrolment may be delayed if, in the opinion of the investigator, the severity of pain represents an isolated incident.
  6. A female subject is eligible to participate if she is of non-childbearing potential.
  7. Body weight <120kg.
  8. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  9. Subject demonstrates an understanding of the study and a willingness to participate as evidenced by voluntary written informed consent.
* Controls:

  1. Subject is either male or female and at least 45 years of age.
  2. Absence of clinically relevant neurologic and psychiatric disease and history of head trauma with loss of consciousness.
  3. Absence of non-compensated medical diseases and pain disorders that may relevantly affect brain function and pain perception.
  4. No clinical evidence of knee OA.
  5. A female subject is eligible to participate if she is of non-childbearing potential.
  6. Body weight <120kg.
  7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  8. Subject demonstrates an understanding of the study and a willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

1. - Subjects will not be permitted to heavily exercise for 12 hours prior to fMRI assessment
2. - Subjects will be required to refrain from the following treatments: I.- Analgesic and anti-inflammatory drugs for 3 days prior to fMRI assessment except for rescue medication. Rescue medication will be based on paracetamol (dosed 1g/8h), which in any case must be withdrawn for a minimum of 24 h prior to fMRI assessment or the fMRI assessment may be delayed.

II.- Steroid injections into the joint or muscle for three months prior to fMRI assessment III.- Hyaluronan injections into index knee within the previous 6 months prior fMRI assessment IV.- Non-pharmacological treatments, such as heat wraps or massage for 24 hours prior to fMRI assessment.

V.- Antidepressants not allowed: MAOIs, Tricyclic antidepressants, mixed 5HT & NE reuptake inhibitors (eg. Duloxetine). SISR are not allowed as a recent prescription, moreover they are allowed in case of chronic use (more than 6 weeks). If those drugs are used for less than 6 weeks, patients could participate in the study after a washout period.

VI.- Anticonvulsant indicated as a pain killer are not allowed, but patients could participate in the study after a washout period.

VII.- Patients can take low doses of hypnotic drugs (eg. Lorazepam 1mg/OD or Diazepam 5mg/OD) if they are used as a chronic prescription (more than 6 weeks). If they are used for less than 6 weeks, patients could participate in the study after a washout period.

Subjects will be allowed to take their chronic (non-analgesic and non-anti-inflammatory) medications if the treatments have been used continuously for at least six weeks prior to assessment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with HIGH / LOW central sensitation, and control subjects.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) in response to pressure stimuli applied to the knee using fMRI | Baseline
  BOLD in response to pressure stimuli applied to the knee assessed using fMRI, that measures endogenous haemodynamic signal reflecting blood oxygenation changes linked to neuronal activity.
BOLD in response to painful contact heat stimuli applied to healthy forearm skin assessed using fMRI | Baseline
  BOLD in response to painful contact heat stimuli applied to healthy forearm skin assessed using fMRI, that measures endogenous haemodynamic signal reflecting blood oxygenation changes linked to neuronal activity.

SECONDARY OUTCOMES:
BOLD during resting-state using fMRI | Baseline
  BOLD during resting-state using fMRI, that measures endogenous haemodynamic signal reflecting blood oxygenation changes linked to neuronal activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Monfort Faure, Barcelona, Barcelona, Spain